CLINICAL TRIAL: NCT01042197
Title: Interdependence Between Body Surface Area and UVB Dose in Vitamin D Production: A Randomized Controlled Trial
Brief Title: The Relation Between Vitamin D Production and UVB Exposed Body Surface Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Vejle Hospital (Other)
Responsible Party: Morten Bogh M.D., Bispebjerg Hospital, Department of Dermatology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H-B-2007-100
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2007-12

CONDITIONS: Vitamin D Status
Keywords: Vitamin D; UVB; Dose-Response; Body surface area

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- 2 (Active Comparator): Body surface area: 12 %
  Interventions: Radiation: Broadband UVB
- 1 (Active Comparator): Body surface area: 6 %
  Interventions: Radiation: Broadband UVB
- 3 (Active Comparator): Body surface area: 24 %
  Interventions: Radiation: Broadband UVB
- 4 (Active Comparator): Body surface area: 6 %
  Interventions: Radiation: Broadband UVB
- 5 (Active Comparator): Body surface area: 12 %
  Interventions: Radiation: Broadband UVB
- 6 (Active Comparator): Body surface area: 24 %
  Interventions: Radiation: Broadband UVB
- 7 (Active Comparator): Body surface area: 6 %
  Interventions: Radiation: Broadband UVB
- 8 (Active Comparator): Body surface area: 12 %
  Interventions: Radiation: Broadband UVB
- 9 (Active Comparator): Body surface area: 24 %
  Interventions: Radiation: Broadband UVB

INTERVENTIONS:
Radiation: Broadband UVB — UVB dose: 0.75 SED. Four UVB sessions with 2 days in between.
  Arms: 1
Radiation: Broadband UVB — UVB dose: 0.75 SED. Four UVB sessions with 2 days in between.
  Arms: 2
Radiation: Broadband UVB — UVB dose: 0.75 SED. Four UVB sessions with 2 days in between.
  Arms: 3
Radiation: Broadband UVB — UVB dose: 1.5 SED. Four UVB sessions with 2 days in between.
  Arms: 4
Radiation: Broadband UVB — UVB dose: 1.5 SED. Four UVB sessions with 2 days in between.
  Arms: 5
Radiation: Broadband UVB — UVB dose: 1.5 SED. Four UVB sessions with 2 days in between.
  Arms: 6
Radiation: Broadband UVB — UVB dose: 3.0 SED. Four UVB sessions with 2 days in between.
  Arms: 7
Radiation: Broadband UVB — UVB dose: 3.0 SED. Four UVB sessions with 2 days in between.
  Arms: 8
Radiation: Broadband UVB — UVB dose: 3.0 SED. Four UVB sessions with 2 days in between.
  Arms: 9

SUMMARY:
The purpose of this study is to investigate the relation between vitamin D production after UVB and exposed body surface areas with different UVB doses.

DETAILED DESCRIPTION:
Vitamin D deficiency is very common. Rachitis, osteoporosis, cancer, sclerosis as well as cardiovascular diseases are related to vitamin D deficiency. Elderly people, immigrants as well as patients with malabsorption diseases often have vitamin D deficiency. 90-95 % of the total vitamin D requirements are obtained from the ultraviolet (UV) radiation of the skin.In spite of the risk of skin-cancer, treatment with sunlight radiation is often recommended against vitamin D deficiency. This fact has raised a scientific debate, where concern has been expressed with regard to the risk of skin-cancer. This dilemma should also be examined as no human studies are available on the vitamin D production in the skin after UV-radiation showing the frequency and dose necessary for sufficient production of vitamin D. The lowest exposure frequency, the smallest body surface area and the lowest UV dose should therefore be established to be exposed in order to minimize the risk of skin-cancer by unnecessary UV-radiation. The purpose of the project is therefore to clarify which factors there are of importance for the production of vitamin D in the skin after UVB radiation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between 18 - 65 years of age.
* Avoidance of sun bed exposure
* Not Holidaying south of 45 degrees latitude 3 months before
* Avoiding vitamin D supplementation during and two months before

Exclusion Criteria:

* Illness as well as age above 65 years.
* Skin diseases
* Psychiatric diseases
* Drug addiction
* Intake of photosensitive medicine.
* Intake of cholesterol-lowering medicine.
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-01; Primary Completion 2009-04 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Vitamin D (nmol/l) measured in a blood sample to define just how much sun exposure is necessary to obtain a sufficient vitamin D production. | Before and 2 days after the last UVB session.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Christian Wulf, Full Prof., Study Chair — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Department of Dermatology D92, Bispebjerg Bakke 23,, Copenhagen Nv, Copenhagen, Denmark